CLINICAL TRIAL: NCT04253509
Title: Clinical Utility of Circulating Tumor DNA Methylation in the Diagnosis of Primary Lung Cancer
Brief Title: Liquid Biopsy Using Methylation Sequencing for Lung Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: EDGC Inc. (Unknown)
Responsible Party: Principal Investigator, Sang-Won Um, Professor, Samsung Medical Center
Other Study IDs: 2019-11-080
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Diagnoses Disease
Keywords: Lung Cancer; Methylation Sequencing; Liquid Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer
  Interventions: Diagnostic Test: Circulating Tumor DNA Methylation Sequencing
- Benign pulmonary disease
  Interventions: Diagnostic Test: Circulating Tumor DNA Methylation Sequencing

INTERVENTIONS:
Diagnostic Test: Circulating Tumor DNA Methylation Sequencing — Whole blood (21mL) collection through venipuncture. Analysis of tumor markers and ctDNA methylation sequencing.

SUMMARY:
This study aims to investigate the utility of circulating tumor DNA (ctDNA) methylation sequencing in the diagnosis of primary lung cancer.

DETAILED DESCRIPTION:
Plasma sample of patients with and without lung cancer will be collected and analyzed using methylation-sensitive enzyme sequencing method. Diagnostic performance of ctDNA methylation sequencing will be compared with that of tumor markers (CEA, Cyfra 21-1, and NSE) combined.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer group

  1. Pathologically proven lung cancer
  2. Clinically suspected lung cancer on chest CT scan
* Benign pulmonary disease group

  * Chronic obstructive pulmonary disease, interstitial lung disease, pneumonia, bronchiectasis, non-tuberculous mycobacterial lung disease, pulmonary vascular disease

Exclusion Criteria:

* Patients with previous history of lung cancer
* Patients who have been diagnosed with other malignancy within 5 years
* Unstable vital status
* Active pulmonary tuberculosis
* Infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Lung cancer
    1. Pathologically proven lung cancer
    2. Clinically suspected lung cancer on chest CT scan
       1. nodule, mass, pulmonary infiltrate, or consolidation
       2. size : diameter at least 1 cm
       3. CT attenuation of solid or part-solid
       4. planned to follow-up, biopsy, or surgical resection
  * Benign pulmonary disease
    1. COPD : post bronchodilator FEV1/FVC < 0.7 and FEV1 pred < 80%
    2. ILD : either histologic or clinical diagnosis
    3. Pneumonia : community or hospital acquired
    4. Bronchiectasis : chest CT diagnosis
    5. NTM : at least 2 isolation of pathogen from sputum
    6. Pulmonary vascular disease : embolism, pulmonary hypertension, arteriovenous malformation
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of ctDNA methylation sequencing | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, diagnostic sensitivity of ctDNA methylation will be compared with that of tumor markers.
Diagnostic specificity of ctDNA methylation sequencing | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, diagnostic specificity of ctDNA methylation will be compared with that of tumor markers.

SECONDARY OUTCOMES:
Diagnostic accuracy of ctDNA methylation sequencing | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, diagnostic accuracy of ctDNA methylation will be compared with that of tumor markers.
Positive predictive value of ctDNA methylation sequencing | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, positive predictive value of ctDNA methylation will be compared with that of tumor markers.
Negative predictive value of ctDNA methylation sequencing | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, negative predictive value of ctDNA methylation will be compared with that of tumor markers.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Won Um, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kwon HJ, Shin SH, Kim HH, Min NY, Lim Y, Joo TW, Lee KJ, Jeong MS, Kim H, Yun SY, Kim Y, Park D, Joo J, Bae JS, Lee S, Jeong BH, Lee K, Lee H, Kim HK, Kim K, Um SW, An C, Lee MS. Advances in methylation analysis of liquid biopsy in early cancer detection of colorectal and lung cancer. Sci Rep. 2023 Aug 19;13(1):13502. doi: 10.1038/s41598-023-40611-w. PMID 37598236